CLINICAL TRIAL: NCT07087132
Title: Translation and Validation of the FS-ICU-24R Into Danish
Status: Recruiting | Type: Observational
Sponsor: Hospitalsenheden Vest (Other)
Collaborators: Aarhus University Hospital (Other); University of Aarhus (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne Højager Nielsen, Head of Research, Hospitalsenheden Vest
Other Study IDs: 1-16-02-51-24
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Family Satisfaction
Keywords: FS-ICU-24R; Intensive Care; Family satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relatives of ICU patients

SUMMARY:
Translation and adaption to a Danish context of the family satisfaction questionnaire FS-ICU-24R. Furthermore, the study will test if the questionnaire adequately measures family satisfaction and is stable over time.

At least 250 relatives of patients, who have been admitted to the intensive care unit at least 24 hours will be included. Relatives will be recruited, when the patients discharge is coming close, i.e. within days. All included relatives will receive the questionnaire on e-mail one month after they registered for the study. Participants will be prompted twice, if they not respond.

After completing the questionnaire once, participants will be asked to complete it a second time after 14 days. The aim is to include at least 50 relatives in this group.

To understand if the questionnaire is measuring family satisfaction, the study will compare the answers to FS-ICU-24R with a score of 1-10 of General satisfaction with the patients care, General satisfaction with information and General satisfaction with decision making. Stability over time will be assessed by comparing responses between first and second time, participants fill out the questionnaire.

Participation will be voluntary and all participants will recieve written and oral information before registering for the study. The participants will register for the study by entering their e-mail into a secure on-line platform.

DETAILED DESCRIPTION:
Method Translation and adaption: The FS-ICU-24R (the family satisfaction with the ICU 24 item questionnarie) will be translated into the Danish language in agreement with one of the original authors, Dr. Daren Heyland. The initial forward translations will be produced by four bilingual nurses all Danish native speakers. Afterwards, the translations will be discussed with two researchers and a pooled version will be produced. Translation of key terms will be thoroughly discussed before deciding on the most appropriate wording. The investigators will opt for a conceptually and culturally sound translation rather than a literal translation, which will be acceptable to the users of the instrument: relatives of ICU patients. Back translation will be undertaken by a bi-lingual nurse, who will be blinded to the original version at all stages of the translation process. The research group will compare the backward version with the source instrument and a second version of the questionnaire will be produced. The process will be repeated to resolve minor discrepancies as needed.

Face and content validity: The Danish version will be presented to 4-6 relatives, who will be interviewed about their perceptions and understanding of the questionnaire. Following the administration of the instrument, all relatives will be interviewed. For each item, relatives will be asked to describe in their own words what they think the item is about and how they chose their answer. Furthermore, if an item is difficult to understand or ambiguous, relatives will be asked to provide alternative wording. Notes and comments made during the interviews on the questionnaire items will be discussed by the researchers before a final version of the questionnaire will be produced. One of the original authors, Dr. Daren Heyland, will approve of the final back translation.

Psychometric testing of FS-ICU-24R in a prospective cohort of Danish ICU relatives:

Recruitment procedure: Relatives will be informed in person about the study while in the ICU. If relatives agree to participate, they must register for the study using a smartphone and a QR code. If a participant prefers to complete the questionnaire on paper, a package containing the questionnaire, information about the study and a return envelope will be supplied with instructions on when to fill in the questionnaire and how to return it. The site will only need to register how many packages have been distributed.

Recruitment of participants to the subgroup test-re-test analysis: When completing the questionnaire in REDCap relatives will be asked to participate a second time for a test-re-test analysis.

Sample size: The reseach group aim to include at least 250 relatives. Several family members from the same family may be included. For criterion and construct validation it is recommended to include more than 100 patients. For confirmatory factor analysis, it is recommended to include 4-10 respondents per item. As the SF-ICU-24R has 26 items and 3 items for bereaved relatives only, at least 250 relatives must be included. Although relatives of the same patient may have some shared experiences, a validation study of the EuroQ2 instrument, which contains many of the same questions, showed that identical ratings only occurred in 28-59% of families. This study supports that relatives' experiences from the same patient trajectory can be surprisingly different. A subgroup of at least 50 relatives will be invited to complete the questionnaire a second time to explore test-retest validity.

Data: In the beginning of the questionnaire, participants will be asked to rate their overall emotional wellbeing, overall satisfaction with care, overall satisfaction with information and overall satisfaction with decision making on Likert scales 1-10 (1= worst imaginable, 10=best imaginable). P participants will then complete the Danish version of the FS-ICU-24R. After each section (satisfaction with care, satisfaction with information, satisfaction with decision making, and bereavement), the participants will be able to make comment in free text. Finally, the participants will be asked to provide background information on sex, age, education, and relationship with the patient.

Data collection: The questionnaire will be distributed by email through the secure web application REDCap hosted by Aarhus University and all data will be stored in REDCap at Aarhus University. For participants preferring to respond in paper, the study group will manually enter mailed responses into REDCap. Paper questionnaires will be coded to identify the issuing ICU.

ELIGIBILITY:
Inclusion Criteria:

* Relative or close friend to an adult patient admitted to the intensive care unit for at least 24 hours.

Exclusion Criteria:

* Persons with cognitive deficits that makes them unable to give informed consent. Persons who cannot read Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relatives to patients admitted to Danish intensive care units.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Family satisfaction | 1 month post discharge from the intensive care unit.
  Summary score of items 1-24 in the FS-ICU-24R questionnaire

OTHER OUTCOMES:
Family satisfaction with care | 1 month post discharge from the intensive care unit.
  Summary score of items 1-14 of the FS-ICU-24R questionnaire
Family satisfaction with decision making | 1 month post discharge from the ICU
  Summary score of the items 15-24 of the FS-ICU-24R questionnaire
Test-retest reliability | one month post ICU discharge
  Spearman's correlation
Construct validity | one month post ICU discharge
  Spearman's correlation
Criterion validity | one month post icu
  The investigators will compare the two subscales with a score of 1-10 of general satisfaction with care, general satisfaction with information and general satisfaction with decision making.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Gødstrup Hospital, Herning

IPD SHARING:
Plan to Share IPD: No
The investigators do not have permission to share data.

REFERENCES:
- [Background] Wall RJ, Engelberg RA, Downey L, Heyland DK, Curtis JR. Refinement, scoring, and validation of the Family Satisfaction in the Intensive Care Unit (FS-ICU) survey. Crit Care Med. 2007 Jan;35(1):271-9. doi: 10.1097/01.CCM.0000251122.15053.50. PMID 17133189
- [Background] Jensen HI, Downey L, Koopmans M, Curtis JR, Engelberg RA, Gerritsen RT. Family ratings of ICU care. Is there concordance within families? J Crit Care. 2020 Feb;55:108-115. doi: 10.1016/j.jcrc.2019.10.011. Epub 2019 Oct 31. PMID 31715527
- [Background] Harrison DA, Ferrando-Vivas P, Wright SE, McColl E, Heyland DK, Rowan KM; Family-Reported Experiences Evaluation Study Investigators. Psychometric assessment of the Family Satisfaction in the Intensive Care Unit questionnaire in the United Kingdom. J Crit Care. 2017 Apr;38:346-350. doi: 10.1016/j.jcrc.2016.10.023. Epub 2016 Nov 5. PMID 27914907
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] De Vet, H. C., Terwee, C. B., Mokkink, L. B., Knol, D. L. (2011). Measurement in medicine : a practical guide. Cambridge University Press.
- [Background] Cha ES, Kim KH, Erlen JA. Translation of scales in cross-cultural research: issues and techniques. J Adv Nurs. 2007 May;58(4):386-95. doi: 10.1111/j.1365-2648.2007.04242.x. Epub 2007 Apr 17. PMID 17442038
- [Derived] Nielsen AH, Agard AS, Collet MO, Brix LD. Translation and Validation of the Canadian ICU Family Satisfaction Questionnaire (FS-ICU-24R) to Danish-A Protocol. Acta Anaesthesiol Scand. 2025 Oct;69(9):e70123. doi: 10.1111/aas.70123. PMID 40922387